CLINICAL TRIAL: NCT02701283
Title: Transcatheter Aortic Valve Replacement With the Medtronic Transcatheter Aortic Valve Replacement System In Patients at Low Risk for Surgical Aortic Valve Replacement
Brief Title: Medtronic Evolut Transcatheter Aortic Valve Replacement in Low Risk Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10234430Doc
Record Dates: First submitted 2016-02-26; First posted 2016-03-08 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Medtronic Transcatheter Aortic Valve Replacement Systems (Experimental): Treatment of Aortic Stenosis with the Medtronic CoreValve System Transcatheter Aortic Valve Implantation (TAVI) device or the Medtronic Corevalve Evolut R System Transcatheter Aortic Valve Implantation (TAVI)
  Interventions: Device: Medtronic Transcatheter Aortic Valve Replacement Systems
- Surgical Aortic Valve Replacement (SAVR) (Active Comparator): Treatment of Aortic Stenosis with commercial Surgical Aortic Valve Replacement (SAVR)
  Interventions: Device: Surgical Aortic Valve Replacement (SAVR)

INTERVENTIONS:
Device: Medtronic Transcatheter Aortic Valve Replacement Systems — Treatment of severe aortic stenosis in subjects who have a low predicted risk of operative mortality for SAVR with Medtronic TAVR Systems
  Arms: Medtronic Transcatheter Aortic Valve Replacement Systems
Device: Surgical Aortic Valve Replacement (SAVR) — Treatment of severe aortic stenosis in subjects who have a low predicted risk of operative mortality for SAVR with a commercially approved surgical bioprothesis
  Arms: Surgical Aortic Valve Replacement (SAVR)

SUMMARY:
The study objective is to demonstrate that the safety and effectiveness of the Medtronic TAVR system as measured by rates of all-cause mortality or disabling stroke at two years is noninferior to SAVR in the treatment of severe aortic stenosis in subjects who have a low predicted risk of operative mortality for SAVR.

The purpose of the expanded use addendum to the Medtronic TAVR in Low Risk Patients Trial protocol is to conclude the randomized phase of the trial and initiate the single-arm, non-randomized, continued access phase of the trial.

DETAILED DESCRIPTION:
Multi-center, international, prospective, randomized, interventional, pre-market.

Subjects will be randomized on 1:1 basis to either TAVR with the Medtronic TAVR system or to SAVR. Patients will be seen at pre and post-procedure, discharge, 30 days, 6 months, 1 year, 18 months, and annually through 10 years.

The expanded use addendum is a multi-center, prospective, non-randomized continued access trial. All heart team approved subjects will be assigned to TAVR with the Medtronic TAVR system. Patients will be seen at pre and post-procedure, discharge, 30 days, and annually through 10 years. Enrollment is expected not to exceed 3660 attempted implants in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic stenosis, defined as follows:

   1. For symptomatic patients:

      Aortic valve area ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), OR mean gradient ≥40 mmHg, OR Maximal aortic valve velocity ≥4.0 m/sec by transthoracic echocardiography at rest
   2. For asymptomatic patients:

      * Very severe aortic stenosis with an aortic valve area of ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), AND maximal aortic velocity ≥5.0 m/sec , or mean gradient ≥60 mmHg by transthoracic echocardiography at rest, OR
      * Aortic valve area of ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), AND a mean gradient ≥40 mmHg or maximal aortic valve velocity ≥4.0 m/sec by transthoracic echocardiography at rest, AND an exercise tolerance test that demonstrates a limited exercise capacity, abnormal BP response, or arrhythmia OR
      * Aortic valve area of ≤1.0 cm2 (or aortic valve area index of ≤0.6 cm2/m2), AND mean gradient ≥40 mmHg, or maximal aortic valve velocity ≥4.0 m/sec by transthoracic echocardiography at rest, AND a left ventricular ejection fraction <50%.
2. Documented heart team agreement of low risk for SAVR, where low risk is defined as predicted risk of mortality for SAVR <3% at 30 days per multidisciplinary local heart team assessment.
3. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

Exclusion Criteria:

1. Any condition considered a contraindication for placement of a bioprosthetic valve (eg, subject is indicated for mechanical prosthetic valve).
2. A known hypersensitivity or contraindication to any of the following that cannot be adequately pre-medicated:

   1. aspirin or heparin (HIT/HITTS) and bivalirudin
   2. ticlopidine and clopidogrel
   3. Nitinol (titanium or nickel)
   4. contrast media
3. Blood dyscrasias as defined: leukopenia (WBC <1000 mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states.
4. Ongoing sepsis, including active endocarditis.
5. Any percutaneous coronary or peripheral interventional procedure with a bare metal stent within 30 days prior to randomization, or drug eluting stent performed within 180 days prior to randomization.
6. Multivessel coronary artery disease with a Syntax score >22 and/or unprotected left main coronary artery.
7. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 10 weeks of Heart Team assessment.
8. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
9. Recent (within 2 months of Heart Team assessment) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
10. Gastrointestinal (GI) bleeding that would preclude anticoagulation.
11. Subject refuses a blood transfusion.
12. Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
13. Estimated life expectancy of less than 24 months due to associated non-cardiac co-morbid conditions.
14. Other medical, social, or psychological conditions that in the opinion of the investigator precludes the subject from appropriate consent or adherence to the protocol required follow-up exams.
15. Currently participating in an investigational drug or another device trial (excluding registries).
16. Evidence of an acute myocardial infarction ≤30 days before the trial procedure due to unstable coronary artery disease (WHO criteria).
17. Need for emergency surgery for any reason.
18. Subject is pregnant or breast feeding.
19. Subject is less than legal age of consent, legally incompetent, or otherwise vulnerable
20. Pre-existing prosthetic heart valve in any position.
21. Severe mitral regurgitation amenable to surgical replacement or repair.
22. Severe tricuspid regurgitation amenable to surgical replacement or repair.
23. Moderate or severe mitral stenosis amenable to surgical replacement or repair.
24. Hypertrophic obstructive cardiomyopathy with left ventricular outflow gradient.
25. Bicuspid aortic valve verified by echocardiography, MDCT, or MRI.
26. Prohibitive left ventricular outflow tract calcification.
27. Sinus of Valsalva diameter unsuitable for placement of the self-expanding bioprosthesis.
28. Aortic annulus diameter of <18 or >30 mm.
29. Significant aortopathy requiring ascending aortic replacement.

    For transfemoral or transaxillary (subclavian) access:
30. Access vessel mean diameter <5.0 mm for Evolut 23R, 26R, or 29R mm TAV, or access vessel mean diameter <5.5 mm for Evolut 34R mm or Evolut PRO TAV. However, for transaxillary (subclavian) access in patients with a patent LIMA, access vessel mean diameter <5.5mm for Evolut 23R, 26R, or 29R mm TAV, or access vessel mean diameter <6.0 mm for the Evolut 34R or Evolut PRO TAV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2223 (Actual)
Dates: Start 2016-03; Primary Completion 2021-04 (Actual); Study Completion 2026-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reardon, MD, Principal Investigator — The Methodist Hospital Research Institute; John K. Forrest, MD, Principal Investigator — Yale New Haven Hospital
Locations (87):
- United States (61):
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - University of Southern California University Hospital, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - Mercy General Hospital, Sacramento, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Morton Plant Hospital, Clearwater, Florida
  - Delray Medical Center, Delray Beach, Florida
  - HealthPark Medical Center, Fort Myers, Florida
  - University of Miami Hospital, Miami, Florida
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Mercy Medical Center, Des Moines, Iowa
  - The University of Kansas Hospital, Kansas City, Kansas
  - Jewish Hospital, Louisville, Kentucky
  - Terrebonne General Medical Center, Houma, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mercy Hospital, Springfield, Missouri
  - Saint Francis Hospital, East Hills, New York
  - Saint Joseph's Hospital Health Center, Liverpool, New York
  - Northwell Health, Manhasset, New York
  - The Mount Sinai Hospital, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Oregon Health Science University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geinsinger Medical Center, Danville, Pennsylvania
  - Pinnacle Health, Harrisburg, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Paramount Heart, Villanova, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Hospital San Antonio, San Antonio, Texas
  - University Hospital Salt Lake City Utah, Salt Lake City, Utah
  - The University of Vermont Medical Center, Burlington, Vermont
  - Saint Mary's Hospital, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Australia (5):
  - Saint Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Monash Health, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital (FSH), Murdoch, Western Australia
- Canada (6):
  - London Health Sciences Centre, London, Ontario
  - Toronto General Health Hospital, Toronto, Ontario
  - Glen Royal Victoria (McGill), Montreal, Quebec
  - IUCPQ, Québec, Quebec
  - Montreal Heart, Montreal
  - Sunnybrook Health Sciences Centre, Toronto
- France (3):
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - L'Hôpital Privé Jacques Cartier Massy, Massy
  - Clinique Pasteur, Toulouse
- Japan (8):
  - Kokura Memorial Hospital, Kitakyushu, Fokuoka
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Teikyo University Hospital, Tokyo, Itabashi-Ku
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - National Cerebral and Cardiovasclular Center, Suita, Osaka
  - The University of Osaka Hospital, Suita, Osaka
  - Sakakibara Heart Institute, Fuchū, Tokyo
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Hospital Nieuwegein, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- Waikato Hospital, Hamilton, New Zealand

REFERENCES:
- [Derived] Erdem S, Goel SS, Reardon MJ. Five-year Outcomes of Transcatheter Aortic Valve Replacement Versus Surgery in Low-risk Aortic Stenosis: Insights from the Evolut Low Risk Trial. Heart Int. 2025 Nov 24;19(2):3-4. doi: 10.17925/HI.2025.19.2.5. eCollection 2025. PMID 41377641
- [Derived] Forrest JK, Yakubov SJ, Deeb GM, Gada H, Mumtaz MA, Ramlawi B, Bajwa T, Crouch J, Merhi W, Wai Sang SL, Kleiman NS, Petrossian G, Robinson NB, Sorajja P, Iskander A, Berthoumieu P, Tchetche D, Feindel C, Horlick EM, Saito S, Oh JK, Jung Y, Reardon MJ; Low Risk Trial Investigators. 5-Year Outcomes After Transcatheter or Surgical Aortic Valve Replacement in Low-Risk Patients With Aortic Stenosis. J Am Coll Cardiol. 2025 Apr 22;85(15):1523-1532. doi: 10.1016/j.jacc.2025.03.004. Epub 2025 Mar 30. PMID 40158212
- [Derived] Butala NM, Lalani C, Tale A, Song Y, Kolte D, Baron S, Strom J, Cohen DJ, Yeh RW. Use of Claims to Assess Outcomes and Treatment Effects in the Evolut Low Risk Trial. Circ Cardiovasc Interv. 2025 Jan;18(1):e014592. doi: 10.1161/CIRCINTERVENTIONS.124.014592. Epub 2025 Jan 21. PMID 39836743
- [Derived] Modine T, Tchetche D, Van Mieghem NM, Deeb GM, Chetcuti SJ, Yakubov SJ, Sorajja P, Gada H, Mumtaz M, Ramlawi B, Bajwa T, Crouch J, Teirstein PS, Kleiman NS, Iskander A, Bagur R, Chu MWA, Berthoumieu P, Sudre A, Adrichem R, Ito S, Huang J, Popma JJ, Forrest JK, Reardon MJ. Three-Year Outcomes Following TAVR in Younger (<75 Years) Low-Surgical-Risk Severe Aortic Stenosis Patients. Circ Cardiovasc Interv. 2024 Nov;17(11):e014018. doi: 10.1161/CIRCINTERVENTIONS.124.014018. Epub 2024 Oct 18. PMID 39421943
- [Derived] Klautz RJM, Rao V, Reardon MJ, Deeb GM, Dagenais F, Moront MG, Little SH, Labrousse L, Patel HJ, Ito S, Li S, Sabik JF 3rd, Oh JK. Examining the typical hemodynamic performance of nearly 3000 modern surgical aortic bioprostheses. Eur J Cardiothorac Surg. 2024 May 3;65(5):ezae122. doi: 10.1093/ejcts/ezae122. PMID 38710669
- [Derived] Tang GHL, Spencer J, Rogers T, Grubb KJ, Gleason P, Gada H, Mahoney P, Dauerman HL, Forrest JK, Reardon MJ, Blanke P, Leipsic JA, Abdel-Wahab M, Attizzani GF, Puri R, Caskey M, Chung CJ, Chen YH, Dudek D, Allen KB, Chhatriwalla AK, Htun WW, Blackman DJ, Tarantini G, Zhingre Sanchez J, Schwartz G, Popma JJ, Sathananthan J. Feasibility of Coronary Access Following Redo-TAVR for Evolut Failure: A Computed Tomography Simulation Study. Circ Cardiovasc Interv. 2023 Nov;16(11):e013238. doi: 10.1161/CIRCINTERVENTIONS.123.013238. Epub 2023 Nov 21. PMID 37988439
- [Derived] Grubb KJ, Shekiladze N, Spencer J, Perdoncin E, Tang GHL, Xie J, Lisko J, Sanchez JZ, Lucas LM, Sathananthan J, Rogers T, Deeb GM, Fukuhara S, Blanke P, Leipsic JA, Forrest JK, Reardon MJ, Gleason P. Feasibility of redo-TAVI in self-expanding Evolut valves: a CT analysis from the Evolut Low Risk Trial substudy. EuroIntervention. 2023 Jul 17;19(4):e330-e339. doi: 10.4244/EIJ-D-22-01125. PMID 37067193
- [Derived] Forrest JK, Deeb GM, Yakubov SJ, Gada H, Mumtaz MA, Ramlawi B, Bajwa T, Teirstein PS, DeFrain M, Muppala M, Rutkin BJ, Chawla A, Jenson B, Chetcuti SJ, Stoler RC, Poulin MF, Khabbaz K, Levack M, Goel K, Tchetche D, Lam KY, Tonino PAL, Ito S, Oh JK, Huang J, Popma JJ, Kleiman N, Reardon MJ; Low Risk Trial Investigators. 3-Year Outcomes After Transcatheter or Surgical Aortic Valve Replacement in Low-Risk Patients With Aortic Stenosis. J Am Coll Cardiol. 2023 May 2;81(17):1663-1674. doi: 10.1016/j.jacc.2023.02.017. Epub 2023 Mar 5. PMID 36882136
- [Derived] Ramlawi B, Deeb GM, Yakubov SJ, Markowitz AH, Hughes GC, Kiaii RB, Huang J, Kleiman NS, Reardon MJ. Mechanisms of Death in Low-Risk Patients After Transcatheter or Surgical Aortic Valve Replacement. Cardiovasc Revasc Med. 2022 Sep;42:1-5. doi: 10.1016/j.carrev.2022.03.027. Epub 2022 Mar 29. PMID 35398007
- [Derived] Forrest JK, Deeb GM, Yakubov SJ, Rovin JD, Mumtaz M, Gada H, O'Hair D, Bajwa T, Sorajja P, Heiser JC, Merhi W, Mangi A, Spriggs DJ, Kleiman NS, Chetcuti SJ, Teirstein PS, Zorn GL 3rd, Tadros P, Tchetche D, Resar JR, Walton A, Gleason TG, Ramlawi B, Iskander A, Caputo R, Oh JK, Huang J, Reardon MJ. 2-Year Outcomes After Transcatheter Versus Surgical Aortic Valve Replacement in Low-Risk Patients. J Am Coll Cardiol. 2022 Mar 8;79(9):882-896. doi: 10.1016/j.jacc.2021.11.062. PMID 35241222
- [Derived] Lanz J, Reardon MJ, Pilgrim T, Stortecky S, Deeb GM, Chetcuti S, Yakubov SJ, Gleason TG, Huang J, Windecker S. Incidence and Outcomes of Infective Endocarditis After Transcatheter or Surgical Aortic Valve Replacement. J Am Heart Assoc. 2021 Oct 5;10(19):e020368. doi: 10.1161/JAHA.120.020368. Epub 2021 Sep 28. PMID 34581194
- [Derived] Blanke P, Leipsic JA, Popma JJ, Yakubov SJ, Deeb GM, Gada H, Mumtaz M, Ramlawi B, Kleiman NS, Sorajja P, Askew J, Meduri CU, Kauten J, Melnitchouk S, Inglessis I, Huang J, Boulware M, Reardon MJ; Evolut Low Risk LTI Substudy Investigators. Bioprosthetic Aortic Valve Leaflet Thickening in the Evolut Low Risk Sub-Study. J Am Coll Cardiol. 2020 May 19;75(19):2430-2442. doi: 10.1016/j.jacc.2020.03.022. Epub 2020 Mar 28. PMID 32234463
- [Derived] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053
- [Derived] Leipsic J, Bax JJ, Webb JG, Martin R, Blanke P. Trials Testing the Value of Imaging Use in Valve Disease and in Transcatheter Valvular Interventions. JACC Cardiovasc Imaging. 2017 Mar;10(3):286-295. doi: 10.1016/j.jcmg.2016.09.031. PMID 28279376

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized Controlled Trial - As Treated
  Continued Access Study - Attempted Implant
Groups:
- Randomized Controlled Trial - Medtronic TAVR Systems: Treatment with Medtronic CoreValve, Evolut R, and Evolut PRO systems in the Randomized Controlled Trial
- Randomized Controlled Trial - SAVR: Surgical Aortic Valve Replacement (SAVR) in the Randomized Controlled Trial
- Continued Access Study - Medtronic TAVR Systems: Treatment with Medtronic Evolut R and Evolut PRO systems in the Continued Access Study
Period: Overall Study
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Started | 737 | 741 | 745
As Treated (Attempted Implant) (Randomized Controlled Trial - The As Treated set includes 4 subjects that crossed over from the Medtronic TAVR Systems arm to the SAVR arm, which accounts for 727 subjects in the Implanted set for the Medtronic TAVR Systems arm. The As Treated set includes 1 subject that crossed over from the SAVR arm to the Medtronic TAVR Systems arm, and 1 subject that was not implanted, which accounts for 686 subjects in the Implanted set for the SAVR arm.) | 730 | 684 | 745
Implanted | 727 | 686 | 745
Completed (The number of completed participants in the Randomized Controlled Trial arms account for the subjects in the As Treated set who completed the 2-year visit. The number of completed participants in the Continued Access Study arm account for the subjects in the Attempted Implant set who completed the 1-year visit.) | 668 | 579 | 724
Not Completed | 69 | 162 | 21
Not completed — Death | 25 | 29 | 19
Not completed — Lost to Follow-up | 3 | 8 | 1
Not completed — Withdrawal by Subject | 12 | 41 | 1
Not completed — Missed 2-year visit | 22 | 27 | 0
Not completed — Exited prior to procedure (3 subjects crossed over from SAVR to TAVR) | 7 | 57 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems | Total
Number analyzed (Participants) | 730 | 684 | 745 | 2159
Age, Continuous [Mean (Standard Deviation); unit: Years] — Subject age reported in years
  Years | 74.1 (5.8) | 73.7 (5.9) | 74.9 (5.9) | 73.9 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266 | 233 | 246 | 745
  Male | 464 | 451 | 499 | 1414
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — Ethnicity was not collected for the Randomized Controlled Trial | NA — Ethnicity was not collected for the Randomized Controlled Trial | 25 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | NA — Ethnicity was not collected for the Randomized Controlled Trial | NA — Ethnicity was not collected for the Randomized Controlled Trial | 705 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Ethnicity was not collected for the Randomized Controlled Trial | NA — Ethnicity was not collected for the Randomized Controlled Trial | 15 | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Race was not collected for the Randomized Controlled Trial | NA — Race was not collected for the Randomized Controlled Trial | 3 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Race was not collected for the Randomized Controlled Trial | NA — Race was not collected for the Randomized Controlled Trial | 4 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Race was not collected for the Randomized Controlled Trial | NA — Race was not collected for the Randomized Controlled Trial | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Race was not collected for the Randomized Controlled Trial | NA — Race was not collected for the Randomized Controlled Trial | 15 | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Race was not collected for the Randomized Controlled Trial | NA — Race was not collected for the Randomized Controlled Trial | 707 | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Race was not collected for the Randomized Controlled Trial | NA — Race was not collected for the Randomized Controlled Trial | 0 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Race was not collected for the Randomized Controlled Trial | NA — Race was not collected for the Randomized Controlled Trial | 15 | NA — Total not calculated because data are not available (NA) in one or more arms.
Subject characteristic - subject age [Mean (Standard Deviation); unit: Years] — Subject age reported in years
  Years | 74.1 (5.8) | 73.7 (5.9) | 74.9 (5.9) | 73.9 (5.9)
Subject characteristic - body surface area [Mean (Standard Deviation); unit: m^2] — Calculated surface area of the human body in m^2
  m^2 | 2.0 (0.2) | 2.0 (0.2) | 2.0 (0.2) | 2.0 (0.2)
Subject characteristic - SYNTAX Score I, Randomized Controlled Trial [Mean (Standard Deviation); unit: Scores on a scale] — SYNTAX Score I is a tool used to calculate the complexity of coronary artery disease Minimum score: 0 Maximum score: 21 Higher values represent more complex coronary artery disease
  Scores on a scale | 1.9 (3.7) | 2.1 (3.9) | NA (NA) — SYNTAX score was not collected for the Continued Access Study | 2.0 (3.8)
Society of Thoracic Surgeons (STS) score [Mean (Standard Deviation); unit: Scores on a scale] — STS score is the of predicted risk of mortality at 30-days Minimum score: 0 Maximum score: 5 Higher values represent a higher risk of mortality at 30-days
  Scores on a scale | 2.0 (0.7) | 1.9 (0.7) | 1.6 (0.6) | 1.9 (0.7)
STS factors [Number; unit: Percent of participants] — Subject characteristics used to calculate STS score
  Percent of participants
    STS Factors Diabetes | 31.4 | 30.7 | 30.4 | 31
    STS Factors Serum Creatinine >2 mg/dl | 0.4 | 0.1 | 0.4 | 0.3
    STS Factors Dialysis | 0.0 | 0.1 | NA — STS Factors Dialysis was not collected for the Continued Access Study | 0.1
    STS Factors Hypertension | 84.8 | 82.4 | 85.0 | 83.6
    STS Factors Endocarditis | 0.0 | 0.0 | 0.0 | 0.0
    STS Factors Chronic Lung Disease (COPD) | 15.1 | 18.0 | 20.3 | 16.5
    STS Factors Immunosuppressive Therapy | 2.1 | 1.0 | 1.1 | 1.6
    STS Factors Peripheral Arterial Disease | 7.5 | 8.2 | 8.7 | 7.8
    STS Factors Cerebrovascular Disease | 10.1 | 12.0 | 2.0 | 11.0
    STS Factors Previous CABG | 2.5 | 2.0 | 2.6 | 2.3
    STS Factors Previous Valve Surgery | 0.0 | 0.0 | 0.0 | 0.0
    STS Factors Previous PCI | 14.1 | 12.9 | 18.3 | 13.5
    STS Factors Previous MI | 6.6 | 4.8 | 8.1 | 5.7
    STS Factors Atrial Fibrillation/ Atrial Flutter | 15.3 | 14.4 | 15.2 | 14.8
New York Heart Association Classification [Number; unit: Percent of participants] — New York Heart Association (NYHA) Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity Class II: Subjects with cardiac disease resulting in slight limitation of physical activity Class III: Subjects with cardiac disease resulting in marked limitation of physical activity Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort
  Percent of participants
    NYHA I | 10.4 | 9.2 | 7.2 | 9.8
    NYHA II | 64.7 | 62.6 | 64.5 | 63.6
    NYHA III | 24.8 | 27.8 | 27.7 | 26.2
    NYHA IV | 0.1 | 0.4 | 0.5 | 0.3
Subject heart conduction disturbances [Number; unit: Percent of participants] — Pre-existing permanent pacemaker or defibrillator: Subject is implanted with a permanent pacemaker or defibrillator at baseline
  Percent of participants | 3.3 | 3.8 | 4.2 | 3.5
Modified Rankin Score (mRS), Randomized Controlled Trial [Number; unit: Percent of participants] — mRS 0: No symptoms mRs 1: No significant disability despite symptoms; able to carry out usual duties and activities.
  mRS 2: Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance.
  mRS 3: Moderate disability; requiring some help, but able to walk without. assistance.
  mRS 4: Moderately severe disability; unable to walk without assistance and unable to attend to own bodily functions.
  mRS 5: Severe disability; bedridden, incontinent and requiring constant nursing care and attention mRS 6: Dead
  Percent of participants
    mRS 0 | 83.8 | 85.0 | NA — mRS was not collected for the Continued Access Study | 84.4
    mRS1 | 9.6 | 8.1 | NA — mRS was not collected for the Continued Access Study | 8.9
    mRS 2 | 5.6 | 6.2 | NA — mRS was not collected for the Continued Access Study | 5.9
    mRS 3 | 1.0 | 0.7 | NA — mRS was not collected for the Continued Access Study | 0.9
    mRS 4 | 0.0 | 0.0 | NA — mRS was not collected for the Continued Access Study | 0.0
    mRS 5 | 0.0 | 0.0 | NA — mRS was not collected for the Continued Access Study | 0.0
    mRS 6 | 0.0 | 0.0 | NA — mRS was not collected for the Continued Access Study | 0.0
Mean aortic gradient [Mean (Standard Deviation); unit: mmHG] — Site reported mean aortic gradient in mmHg recorded at baseline
  mmHG | 46.9 (12.2) | 46.5 (12.2) | 45.5 (12.5) | 46.7 (12.2)
Max aortic valve velocity [Mean (Standard Deviation); unit: m/sec] — Site reported maximum aortic valve velocity measured in m/sec
  m/sec | 4.4 (0.5) | 4.4 (0.5) | 4.3 (0.5) | 4.4 (0.5)
Aortic valve area (AVA) [Mean (Standard Deviation); unit: cm2] — Site reported aortic valve area measured in cm^2
  cm2 | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.2)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: Percentage of blood ejected] — Site reported LVEF measured is the percent of the blood ejected by the left ventricle when contracting
  Percentage of blood ejected | 61.7 (7.9) | 61.9 (7.7) | 61.8 (8.0) | 61.8 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Safety: All Cause Mortality or Disabling Stroke Rate at 24 Months, Randomized Controlled Trial Safety: All Cause Mortality or All Stroke Rate at 12 Months, Continued Access Study
Description: Assessment of procedural safety by:
  All-cause mortality: all deaths from any cause after valve intervention. This includes all cardiovascular and non-cardiovascular deaths.
  Disabling stroke: a modified rankin score (mRS) of 2 or more at 90 days post-stroke and an increase of at least one mRS category from an individual's pre-stroke baseline.
  All stroke: any stroke after valve intervention (ischemic, hemorrhagic, or undetermined stroke).
Time Frame: Randomized Controlled Trial - 24 months Continued Access Study - 12 months
Population: Randomized Controlled Trial - As treated set Continued Access Study - Attempted implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 730 | 684 | 745
Percent of participants (K-M rate) | 4.3 | 6.3 | 5.7
Statistical Analysis 1: Comparison: Randomized Controlled Trial - Medtronic TAVR Systems vs Randomized Controlled Trial - SAVR; Primary Hypothesis: TAVR with the Medtronic TAVR system is non-inferior to SAVR for all-cause mortality or disabling stroke rate during a fixed follow-up of 24 months for the Randomized Controlled Trial; Test type: Non-Inferiority — Absolute non-inferiority margin was 0.06; Bayesian — The posterior probability of non-inferiority is > 0.999. The posterior probability is the probability of the event rate by updating the prior probability distribution with observed data at the interim analysis using Bayes' Theorem; Posterior Median of the Difference = 0.999 — 95% Bayesian credible interval for the difference (TAVR-SAVR) was (-4.4%, 0.4%). The 95% credible interval is the 2.5th and 97.5th percentiles of the posterior distribution

2. Secondary Outcome: RCT: Composite of Death, Disabling Stroke, Life-threatening Bleed, Major Vascular Complication, or AKI (II or III) at 30 Days CAS: Composite of Death, All Stroke, Life-threatening Bleed, or Major Vascular Complication at 30 Days
Description: Randomized Controlled Trial: Combined clinical efficacy after 30 days was defined as the composite of all-cause mortality, disabling stroke, life-threatening bleed, major vascular complication, or AKI (II or III)
  Continued Access Study: Combined clinical efficacy after 30 days was defined as the composite of all-cause mortality, all stroke, life-threatening bleed, or major vascular complication
Time Frame: 30 days
Population: As treated set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 730 | 684 | 745
Percent of participants (K-M rate)
  Composite event | 5.3 | 10.8 | 6.6
  Death | 0.4 | 1.2 | 0.7
  Disabling stroke | 0.4 | 1.6 | NA — The 30 day composite endpoint for the Continued Access Study included all strokes, not disabling strokes separately.
  Life-threatening or disabling bleed | 2.5 | 7.5 | 3.4
  Major vascular complication | 3.7 | 3.1 | 0.4
  AKI (II or III) | 0.8 | 2.8 | NA — AKI (II or III) was not assessed for the Continued Access Study
  All Stroke | NA — The 30 day composite endpoint for the Randomized Controlled Trial included disabling strokes, not all strokes as a component. | NA — The 30 day composite endpoint for the Randomized Controlled Trial included disabling strokes, not all strokes as a component. | 2.7

3. Secondary Outcome: New Pacemaker Implantation at 30 Days
Description: The rate of new permanent pacemaker implant at 30 days
Time Frame: 30 days
Population: Randomized Controlled Trial - As treated set Continued Access Study - Attempted implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 730 | 684 | 745
Percent of participants (K-M rate) | 17.7 | 6.3 | 15.0

4. Secondary Outcome: Prosthetic Valve Endocarditis at 1 Year
Description: The rate of prosthetic valve endocarditis at 1 year
Time Frame: 1 year
Population: Randomized Controlled Trial - As treated set Continued Access Study - Attempted implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 730 | 684 | 745
Percent of participants (K-M rate) | 0.1 | 0.5 | 0.4

5. Secondary Outcome: Prosthetic Valve Thrombosis at 1 Year
Description: The rate of prosthetic valve thrombosis at 1 year
Time Frame: 1 year
Population: Randomized Controlled Trial - As treated set Continued Access Study - Attempted implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 730 | 684 | 745
Percent of participants (K-M rate) | 0.3 | 0.2 | 0.0

6. Secondary Outcome: All Stroke (Disabling and Non-disabling) at 1 Year
Description: The rate of all stroke (disabling and non-disabling) at 1 year
Time Frame: 1 year
Population: Randomized Controlled Trial - As treated set Continued Access Study - Attempted implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 730 | 684 | 745
Percent of participants (K-M rate) | 4.3 | 4.3 | 3.6

7. Secondary Outcome: Life-threatening Bleeding at 1 Year
Description: The rate of life-threatening bleeding at 1 year
Time Frame: 1 year
Population: Randomized Controlled Trial - As treated set Continued Access Study - Attempted implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 730 | 684 | 745
Percent of participants (K-M rate) | 3.6 | 8.7 | 3.8

8. Secondary Outcome: Valve-related Dysfunction Requiring Repeat Procedure at 1 Year
Description: The rate of valve-related dysfunction requiring repeat procedure at 1 year
Time Frame: 1 year
Population: Randomized Controlled Trial - As treated set Continued Access Study - Attempted implant set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 730 | 684 | 745
Percent of participants (K-M rate) | 0.6 | 0.4 | 0.8

9. Secondary Outcome: Valve-related Dysfunction (Moderate or Severe Stenosis or Regurgitation) at 1 Year, Randomized Controlled Trial
Description: Stenosis (moderate or severe)
  Any of the following:
  1. Peak aortic velocity >4 m/s OR mean aortic gradient >40 mmHg, AND EOA <0.8 cm2
  2. Peak aortic velocity >4 m/s OR mean aortic gradient >40 mmHg, AND EOA ≥0.8 cm2, and DVI <0.25
  3. Peak aortic velocity ≤4 m/s and mean aortic gradient ≤ 40 mmHg, AND EOA <0.8 cm2, and DVI <0.25
  Regurgitation (moderate or severe)
  Any of the following:
  1. Moderate or Severe Total Regurgitation
  2. Moderate or Severe Paravalvular Regurgitation
  3. Moderate or Severe Transvalvular Regurgitation
Time Frame: 1 year
Population: Implanted
Measure: Number; unit: Percent of participants
Groups:
- Medtronic TAVR Systems: Treatment with Medtronic CoreValve, Evolut R, and Evolut PRO systems
- SAVR: Surgical Aortic Valve Replacement (SAVR)
Arm/Group | Medtronic TAVR Systems | SAVR
Number analyzed (Participants) | 727 | 686
Percent of participants
  Moderate or severe stenosis | 0.2 | 0.4
  Moderate or severe regurgitation | 4.3 | 1.3

10. Secondary Outcome: Randomized Controlled Trial - Health-related Quality of Life as Assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) at 30 Days and 1 Year Continued Access Study - Health-related Quality of Life as Assessed by KCCQ at 1 Year
Description: Quality of life summary scores and change from baseline using the following measures:
  KCCQ: Quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Randomized Controlled Trial - 30 days and 1 year Continued Access Study - 1 year
Population: Randomized Controlled Trial - As treated set Continued Access Study - Attempted implant set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 730 | 684 | 745
Score on a scale
  30 day KCCQ - Overall | 88.6 (14.2) | 78.7 (18.8) | NA (NA) — 30 day KCCQ scores were not an endpoint measure for the Continued Access Study
  30 day change from baseline - Overall | 20.0 (21.1) | 9.2 (22.3) | NA (NA) — 30 day KCCQ scores were not an endpoint measure for the Continued Access Study
  30 day KCCQ - Clinical | 89.7 (13.4) | 82.6 (16.9) | NA (NA) — 30 day KCCQ scores were not an endpoint measure for the Continued Access Study
  30 day change from baseline - Clinical | 15.4 (19.6) | 7.5 (20.5) | NA (NA) — 30 day KCCQ scores were not an endpoint measure for the Continued Access Study
  1 year KCCQ - Overall | 90.6 (12.7) | 90.5 (12.4) | 91.1 (13.8)
  1 year change from baseline - Overall | 21.6 (20.6) | 20.7 (20.3) | 24.7 (22.8)
  1 year KCCQ - Clinical | 89.9 (13.4) | 90.2 (12.8) | NA (NA) — KCCQ Clinical score was not calculated for the Continued Access Study
  1 year change from baseline - Clinical | 15.3 (18.9) | 14.8 (18.9) | NA (NA) — KCCQ Clinical score was not calculated for the Continued Access Study

11. Secondary Outcome: Repeat Hospitalization for Aortic Valve Disease at 1 Year, Randomized Controlled Trial
Description: The rate of repeat hospitalization for aortic valve disease at 1 year
Time Frame: 1 year
Population: As treated set
Measure: Number; unit: Percent of participants (K-M rate)
Arm/Group | Medtronic TAVR Systems | SAVR
Number analyzed (Participants) | 730 | 684
Percent of participants (K-M rate) | 3.5 | 5.8

12. Other Pre Specified Outcome: Hemodynamic Performance Metrics by Doppler Echocardiography: Percent of Participants With Degrees of Total Prosthetic Valve Regurgitation at 1 Year, Randomized Controlled Trial
Description: Reporting of prosthetic valve hemodynamic performance by degree of total prosthetic valve regurgitation
Time Frame: 1 year
Population: Implanted
Measure: Number; unit: Percent of participants
Arm/Group | Medtronic TAVR Systems | SAVR
Number analyzed (Participants) | 727 | 686
Percent of participants
  None | 39.4 | 72.2
  Trace | 23.5 | 19.3
  Mild/Mild to Moderate | 32.9 | 7.2
  Moderate/Moderate to Severe | 4.1 | 1.3
  Severe | 0.1 | 0.0

13. Other Pre Specified Outcome: Hemodynamic Performance Metrics by Doppler Echocardiography at 1 Year, Randomized Controlled Trial Effective Orifice Area (EOA) at 1 Year
Description: Reporting of prosthetic valve hemodynamic performance by EOA
Time Frame: 1 year
Population: Implanted
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Medtronic TAVR Systems | SAVR
Number analyzed (Participants) | 727 | 686
cm2 | 2.23 (0.63) | 1.96 (0.57)

14. Other Pre Specified Outcome: Health-related Quality of Life as Assessed by European QoL (EQ-5D) at 1 Year, Randomized Controlled Trial
Description: Quality of life summary scores and change from baseline using the following measures:
  EQ-5D: Measures 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that can be converted to utilities using an algorithm. Utilities range from 0 to 1, with 1 representing perfect health, and 0 corresponding to the worst imaginable health state
Time Frame: 1 year
Population: As treated set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Medtronic TAVR Systems | SAVR
Number analyzed (Participants) | 730 | 684
Score on a scale
  EQ-5D Index Score at 1 year | 0.81 (0.21) | 0.81 (0.19)
  1 year change from baseline EQ-5D Index Score | 0.09 (0.24) | 0.08 (0.24)

15. Other Pre Specified Outcome: New York Heart Association (NYHA) Functional Classification at 1 Year, Randomized Controlled Trial
Description: Reporting of NYHA classification at 1 year
  NYHA Classification criteria:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity Class I: Subjects with cardiac disease resulting in slight limitation of physical activity Class III: Subjects with cardiac disease resulting in marked limitation of physical activity Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort
Time Frame: 1 year
Population: As treated set
Measure: Number; unit: Percent of participants
Arm/Group | Medtronic TAVR Systems | SAVR
Number analyzed (Participants) | 730 | 684
Percent of participants
  NYHA Class I | 80.6 | 79.5
  NYHA Class II | 15.8 | 15.7
  NYHA Class III | 1.1 | 1.4
  NYHA Class IV | 0.4 | 0.3
  Died prior to visit | 2.1 | 3.0

16. Other Pre Specified Outcome: Hemodynamic Performance Metrics by Doppler Echocardiography at 1 Year, Randomized Controlled Trial Mean Aortic Gradient at 1 Year
Description: Reporting of prosthetic valve hemodynamic performance by transvalvular mean aortic gradient
Time Frame: 1 year
Population: Implanted
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Medtronic TAVR Systems | SAVR
Number analyzed (Participants) | 727 | 686
mmHG | 8.74 (3.58) | 11.27 (4.81)

17. Other Pre Specified Outcome: Efficacy: Device Success Rate
Description: Assessment of procedural effectiveness by meeting all of the following device success criteria:
  * Absence of procedural mortality, AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location, AND
  * Absence of moderate or severe total prosthetic valve regurgitation (at 18 hours to 7 days)
Time Frame: Hospital discharge or 7 days post-procedure (whichever occurs first)
Population: Randomized Controlled Trial - Implanted set. Per the Clinical Investigational Plan, the incidence estimate is provided for the TAVR group only.
  Continued Access Study - Attempted implant set.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Continued Access Study - Medtronic TAVR Systems
Number analyzed (Participants) | 727 | 745
Percent of participants | 85.3 [82.1 to 88.1] | 98.1 [96.9 to 99]

ADVERSE EVENTS:
Time Frame: Randomized Controlled Trial - Adverse events (AEs) were collected from study enrollment through the 24 month follow-up visit. Adverse event data are currently available and reported for up to 24 months. Continued Access Study - Adverse events (AEs) were collected from study enrollment through the 12 month follow-up visit. Adverse event data are currently available and reported for up to 12 months.
Description: Randomized Controlled Trial - All new or worsening AEs were collected through 24 months. After 24 months only serious and device-related events will be collected.
  Continued Access Study - All new or worsening AEs were collected through 12 months. Note, any AE that is entered as 0 for this portion of the study does not imply that the AE did not occur, rather it is not collected in the TVT Registry. There are no events entered in the 'Other' table as TVT-R does not distinguish seriousness.
Arm/Group | Randomized Controlled Trial - Medtronic TAVR Systems | Randomized Controlled Trial - SAVR | Continued Access Study - Medtronic TAVR Systems
All-Cause Mortality (participants affected / at risk) | 25/730 | 29/684 | 19/745
Serious Adverse Events (participants affected / at risk) | 459/730 | 495/684 | 429/745
Other Adverse Events (participants affected / at risk) | 474/730 | 571/684 | 0/745
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Controlled Trial - Medtronic TAVR Systems (N=730) | Randomized Controlled Trial - SAVR (N=684) | Continued Access Study - Medtronic TAVR Systems (N=745)
Anaemia (Blood and lymphatic system disorders) | 22 | 60 | 0
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 | 21 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 7 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Hypergammaglobulinaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 27 | 0
Acquired Cardiac Septal Defect (Cardiac disorders) | 0 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 1 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 3 | 2 | 0
Acute Myocardial Infarction (Cardiac disorders) | 8 | 5 | 4
Angina Pectoris (Cardiac disorders) | 2 | 3 | 0
Angina Unstable (Cardiac disorders) | 0 | 1 | 0
Aortic Valve Calcification (Cardiac disorders) | 0 | 1 | 0
Aortic Valve Incompetence (Cardiac disorders) | 6 | 2 | 0
Aortic Valve Stenosis (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 3 | 1 | 0
Arteriospasm Coronary (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 38 | 135 | 12
Atrial Flutter (Cardiac disorders) | 6 | 20 | 0
Atrial Tachycardia (Cardiac disorders) | 1 | 1 | 0
Atrial Thrombosis (Cardiac disorders) | 0 | 2 | 0
Atrioventricular Block (Cardiac disorders) | 2 | 2 | 0
Atrioventricular Block Complete (Cardiac disorders) | 89 | 36 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 12 | 1 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 13 | 5 | 0
Atrioventricular Dissociation (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 9 | 5 | 0
Bundle Branch Block Left (Cardiac disorders) | 29 | 3 | 0
Bundle Branch Block Right (Cardiac disorders) | 3 | 1 | 0
Cardiac Amyloidosis (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 11 | 11 | 7
Cardiac Failure (Cardiac disorders) | 4 | 5 | 0
Cardiac Failure Acute (Cardiac disorders) | 3 | 2 | 0
Cardiac Failure Chronic (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 16 | 24 | 0
Cardiac Tamponade (Cardiac disorders) | 1 | 3 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 2 | 2 | 0
Cardiogenic Shock (Cardiac disorders) | 4 | 6 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 0
Cardiopulmonary Failure (Cardiac disorders) | 2 | 0 | 0
Conduction Disorder (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 4 | 3 | 0
Coronary Artery Dissection (Cardiac disorders) | 0 | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 6 | 3 | 0
Coronary Ostial Stenosis (Cardiac disorders) | 0 | 1 | 0
Diastolic Dysfunction (Cardiac disorders) | 1 | 0 | 0
Dressler's Syndrome (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 2 | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 1 | 2 | 0
Left Ventricular Hypertrophy (Cardiac disorders) | 0 | 1 | 0
Low Cardiac Output Syndrome (Cardiac disorders) | 0 | 2 | 0
Mitral Valve Incompetence (Cardiac disorders) | 2 | 3 | 0
Myocardial Haemorrhage (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 2 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 2 | 0
Nodal Rhythm (Cardiac disorders) | 1 | 4 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Paroxysmal Atrioventricular Block (Cardiac disorders) | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 8 | 9 | 0
Pericardial Haemorrhage (Cardiac disorders) | 1 | 5 | 0
Pericarditis (Cardiac disorders) | 3 | 0 | 0
Pleuropericarditis (Cardiac disorders) | 0 | 1 | 0
Prosthetic Cardiac Valve Thrombosis (Cardiac disorders) | 1 | 3 | 0
Pulseless Electrical Activity (Cardiac disorders) | 0 | 2 | 0
Right Ventricular Dysfunction (Cardiac disorders) | 0 | 1 | 0
Sinus Arrest (Cardiac disorders) | 2 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 3 | 2 | 0
Sinus Node Dysfunction (Cardiac disorders) | 10 | 8 | 0
Supraventricular Tachycardia (Cardiac disorders) | 2 | 7 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 2 | 3 | 0
Ventricular Fibrillation (Cardiac disorders) | 6 | 6 | 0
Ventricular Tachycardia (Cardiac disorders) | 9 | 7 | 0
Hypertrophic Cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 2 | 0
Meniere's Disease (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 0
Adrenal Mass (Endocrine disorders) | 1 | 0 | 0
Thyroid Mass (Endocrine disorders) | 1 | 1 | 0
Blindness (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 8 | 3 | 0
Cataract Nuclear (Eye disorders) | 0 | 1 | 0
Corneal Degeneration (Eye disorders) | 1 | 0 | 0
Macular Hole (Eye disorders) | 0 | 1 | 0
Macular Oedema (Eye disorders) | 1 | 0 | 0
Optic Ischaemic Neuropathy (Eye disorders) | 0 | 1 | 0
Retinal Artery Occlusion (Eye disorders) | 1 | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 2 | 0
Retinal Vein Occlusion (Eye disorders) | 1 | 0 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 1 | 0
Visual Impairment (Eye disorders) | 1 | 1 | 0
Vitreous Haemorrhage (Eye disorders) | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 3 | 0
Abdominal Mass (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Acquired Oesophageal Web (Gastrointestinal disorders) | 0 | 1 | 0
Appendiceal Mucocoele (Gastrointestinal disorders) | 0 | 1 | 0
Barrett's Oesophagus (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 6 | 0
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Faeces Discoloured (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Polyps (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Angiectasia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 11 | 5 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2 | 0
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 | 2 | 0
Inguinal Hernia (Gastrointestinal disorders) | 6 | 2 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 2 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 1 | 0
Mesenteritis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 0
Obstructive Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Oesophageal Motility Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 4 | 0
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 3 | 3 | 0
Retroperitoneal Haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 3 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 3 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Asthenia (General disorders) | 0 | 4 | 0
Chest Discomfort (General disorders) | 2 | 0 | 0
Chest Pain (General disorders) | 11 | 11 | 0
Critical Illness (General disorders) | 0 | 1 | 0
Death (General disorders) | 2 | 3 | 19
Device Embolisation (General disorders) | 1 | 0 | 2
Extravasation (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0
Generalised Oedema (General disorders) | 0 | 2 | 0
Granuloma (General disorders) | 0 | 1 | 0
Hernia (General disorders) | 0 | 1 | 0
Infusion Site Extravasation (General disorders) | 0 | 2 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 3 | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 2 | 0
Oedema (General disorders) | 0 | 2 | 0
Oedema Peripheral (General disorders) | 3 | 1 | 0
Pain (General disorders) | 1 | 1 | 0
Pelvic Mass (General disorders) | 0 | 1 | 0
Polyp (General disorders) | 1 | 0 | 0
Puncture Site Haemorrhage (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 8 | 6 | 0
Stent-Graft Endoleak (General disorders) | 0 | 1 | 0
Swelling (General disorders) | 1 | 0 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 2 | 0
Vascular Stent Stenosis (General disorders) | 0 | 1 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 0 | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 4 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 5 | 0
Gallbladder Fistula (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 2 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 0 | 1 | 0
Ischaemic Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 1 | 0
Arthritis Infective (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 3 | 4 | 0
Bartholin's Abscess (Infections and infestations) | 0 | 1 | 0
Biliary Sepsis (Infections and infestations) | 1 | 1 | 0
Brain Abscess (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 3 | 0
Cardiac Valve Abscess (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 8 | 10 | 0
Chronic Sinusitis (Infections and infestations) | 1 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 4 | 0
Coccidioidomycosis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Device Related Infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 0
Endocarditis (Infections and infestations) | 3 | 6 | 3
Enterococcal Infection (Infections and infestations) | 0 | 1 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 0
Groin Abscess (Infections and infestations) | 1 | 0 | 0
Implant Site Infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 2 | 1 | 0
Influenza (Infections and infestations) | 5 | 2 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Lyme Disease (Infections and infestations) | 0 | 1 | 0
Mediastinitis (Infections and infestations) | 0 | 2 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis Bacterial (Infections and infestations) | 0 | 1 | 0
Otitis Media (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 11 | 28 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 4 | 0
Pseudomonas Bronchitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 8 | 13 | 0
Septic Shock (Infections and infestations) | 1 | 6 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin Graft Infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 2 | 1 | 0
Streptococcal Bacteraemia (Infections and infestations) | 1 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 16 | 10 | 0
Urosepsis (Infections and infestations) | 2 | 2 | 0
Vascular Access Site Infection (Infections and infestations) | 0 | 1 | 0
Wound Infection (Infections and infestations) | 1 | 4 | 0
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 | 20 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Aortic Injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Arterial Injury (Injury, poisoning and procedural complications) | 3 | 0 | 0
Cardiac Valve Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Central Nervous System Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 6 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Foreign Body (Injury, poisoning and procedural complications) | 1 | 1 | 0
Foreign Body In Gastrointestinal Tract (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heart Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 8 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision Site Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 3 | 0 | 0
Metaphyseal Corner Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Periprocedural Myocardial Infarction (Injury, poisoning and procedural complications) | 1 | 3 | 0
Phrenic Nerve Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Fever (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 6 | 0
Post Procedural Hypotension (Injury, poisoning and procedural complications) | 0 | 2 | 0
Postoperative Delirium (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative Hypertension (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 0 | 2 | 0
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postpericardiotomy Syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 19 | 0
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation Proctitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation Retinopathy (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 1 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 3 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 3 | 2 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Suture Related Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urethral Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular Access Site Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular Access Site Dissection (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 2
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 7
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 4 | 2 | 0
Vasoplegia Syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 3 | 0
Wound Secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anticoagulation Drug Level Above Therapeutic (Investigations) | 0 | 3 | 0
Blood Creatinine Increased (Investigations) | 0 | 1 | 0
Blood Magnesium Decreased (Investigations) | 0 | 1 | 0
Brain Natriuretic Peptide Increased (Investigations) | 1 | 0 | 0
C-Reactive Protein Increased (Investigations) | 1 | 0 | 0
Cardiac Output Decreased (Investigations) | 0 | 1 | 0
Computerised Tomogram Abnormal (Investigations) | 1 | 0 | 0
Echocardiogram Abnormal (Investigations) | 1 | 0 | 0
Ejection Fraction Decreased (Investigations) | 1 | 2 | 0
Electrocardiogram Qrs Complex Prolonged (Investigations) | 0 | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 2 | 0
Heart Rate Irregular (Investigations) | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 1 | 0
Mammogram Abnormal (Investigations) | 0 | 1 | 0
Occult Blood (Investigations) | 0 | 1 | 0
Red Blood Cell Analysis Abnormal (Investigations) | 0 | 1 | 0
Transvalvular Pressure Gradient Increased (Investigations) | 1 | 0 | 0
Troponin Increased (Investigations) | 2 | 0 | 0
Urine Output Decreased (Investigations) | 0 | 5 | 0
Vascular Resistance Systemic (Investigations) | 0 | 1 | 0
Wall Motion Score Index Abnormal (Investigations) | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Body Fat Disorder (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 5 | 0
Failure To Thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 5 | 29 | 0
Gout (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 18 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 5 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 10 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 11 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 6 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 11 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 6 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 4 | 0
Lactic Acidosis (Metabolism and nutrition disorders) | 1 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 3 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 3 | 0
Metabolic Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Chest Wall Haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral Disc Displacement (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 | 11 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenoid Cystic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
High-Grade B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant Neoplasm Of Renal Pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Nasal Sinus Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 0
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Altered State Of Consciousness (Nervous system disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 2 | 1 | 0
Brain Injury (Nervous system disorders) | 2 | 1 | 0
Brain Stem Stroke (Nervous system disorders) | 1 | 0 | 0
Carotid Artery Disease (Nervous system disorders) | 1 | 0 | 0
Carotid Artery Occlusion (Nervous system disorders) | 1 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 5 | 2 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 5 | 1 | 0
Cerebral Haematoma (Nervous system disorders) | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 2 | 2 | 0
Cerebral Small Vessel Ischaemic Disease (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 19 | 23 | 4
Cervical Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Dementia With Lewy Bodies (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 4 | 0
Dysarthria (Nervous system disorders) | 2 | 0 | 0
Embolic Stroke (Nervous system disorders) | 2 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 7 | 0
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 2 | 3 | 0
Hemianopia (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 2 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Hypercapnic Coma (Nervous system disorders) | 0 | 1 | 0
Hypertensive Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypokinesia (Nervous system disorders) | 0 | 1 | 0
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Intracranial Hypotension (Nervous system disorders) | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 4 | 3 | 25
Lumbar Radiculopathy (Nervous system disorders) | 3 | 1 | 0
Lumbosacral Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Metabolic Encephalopathy (Nervous system disorders) | 1 | 2 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0
Neuromyopathy (Nervous system disorders) | 1 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 2 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Postictal State (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 4 | 0
Seizure (Nervous system disorders) | 2 | 4 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 18 | 7 | 0
Tarsal Tunnel Syndrome (Nervous system disorders) | 1 | 0 | 0
Tension Headache (Nervous system disorders) | 1 | 0 | 0
Thalamic Infarction (Nervous system disorders) | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 12 | 9 | 5
Trigeminal Neuralgia (Nervous system disorders) | 1 | 0 | 0
Vascular Dementia (Nervous system disorders) | 0 | 1 | 0
Device Breakage (Product Issues) | 0 | 1 | 0
Device Dislocation (Product Issues) | 3 | 0 | 1
Device Failure (Product Issues) | 0 | 1 | 0
Device Leakage (Product Issues) | 3 | 3 | 0
Device Loosening (Product Issues) | 0 | 1 | 0
Device Physical Property Issue (Product Issues) | 1 | 0 | 0
Lead Dislodgement (Product Issues) | 2 | 1 | 0
Thrombosis In Device (Product Issues) | 0 | 1 | 0
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Completed Suicide (Psychiatric disorders) | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 2 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0
Delirium Tremens (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 12 | 27 | 0
Bladder Mass (Renal and urinary disorders) | 1 | 0 | 0
Bladder Outlet Obstruction (Renal and urinary disorders) | 1 | 0 | 0
Calculus Bladder (Renal and urinary disorders) | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 9 | 4 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 3 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 1 | 0
Renal Cyst (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 5 | 7 | 0
Subcapsular Renal Haematoma (Renal and urinary disorders) | 0 | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 11 | 12 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2 | 1 | 0
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular Pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 0
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Mediastinal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 49 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 10 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 10 | 27 | 0
Thoracic Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ischaemic Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pyoderma Gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aneurysm Repair (Surgical and medical procedures) | 1 | 0 | 0
Ankle Operation (Surgical and medical procedures) | 1 | 0 | 0
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 1 | 0 | 110
Carpal Tunnel Decompression (Surgical and medical procedures) | 1 | 1 | 0
Cataract Operation (Surgical and medical procedures) | 2 | 1 | 0
Coronary Endarterectomy (Surgical and medical procedures) | 0 | 1 | 0
Drain Removal (Surgical and medical procedures) | 0 | 1 | 0
Hernia Repair (Surgical and medical procedures) | 1 | 1 | 0
Hip Arthroplasty (Surgical and medical procedures) | 3 | 1 | 0
Hip Surgery (Surgical and medical procedures) | 1 | 0 | 0
Knee Arthroplasty (Surgical and medical procedures) | 5 | 2 | 0
Shoulder Arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Spinal Fusion Surgery (Surgical and medical procedures) | 1 | 0 | 0
Thoracic Cavity Drainage (Surgical and medical procedures) | 0 | 2 | 0
Toe Amputation (Surgical and medical procedures) | 2 | 0 | 0
Tooth Extraction (Surgical and medical procedures) | 1 | 0 | 0
Transurethral Bladder Resection (Surgical and medical procedures) | 2 | 0 | 0
Angiopathy (Vascular disorders) | 2 | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 1 | 0
Aortic Arteriosclerosis (Vascular disorders) | 0 | 2 | 0
Aortic Dissection (Vascular disorders) | 1 | 1 | 0
Aortic Perforation (Vascular disorders) | 0 | 1 | 0
Aortic Stenosis (Vascular disorders) | 1 | 0 | 0
Aortic Thrombosis (Vascular disorders) | 1 | 1 | 0
Arterial Haemorrhage (Vascular disorders) | 1 | 0 | 0
Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0
Arterial Thrombosis (Vascular disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Artery Dissection (Vascular disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 5 | 0
Femoral Artery Aneurysm (Vascular disorders) | 1 | 0 | 0
Femoral Artery Dissection (Vascular disorders) | 3 | 0 | 0
Haematoma (Vascular disorders) | 7 | 3 | 0
Haemodynamic Instability (Vascular disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 6 | 4 | 18
Hypertension (Vascular disorders) | 13 | 33 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 1 | 0
Hypertensive Urgency (Vascular disorders) | 3 | 0 | 0
Hypotension (Vascular disorders) | 39 | 38 | 0
Hypovolaemic Shock (Vascular disorders) | 0 | 1 | 0
Intermittent Claudication (Vascular disorders) | 2 | 0 | 0
Lymphorrhoea (Vascular disorders) | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 10 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 3 | 2 | 0
Peripheral Artery Dissection (Vascular disorders) | 5 | 0 | 0
Peripheral Artery Occlusion (Vascular disorders) | 2 | 0 | 0
Peripheral Artery Stenosis (Vascular disorders) | 2 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 2 | 0 | 0
Peripheral Venous Disease (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 3 | 0
Shock Haemorrhagic (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 2 | 0
Thrombosis (Vascular disorders) | 2 | 1 | 0
Vasodilatation (Vascular disorders) | 0 | 1 | 0
Coronary artery compression (Cardiac disorders) | 0 | 0 | 1
Complication associated with device (General disorders) | 0 | 0 | 7
Perforation (General disorders) | 0 | 0 | 4
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 | 0 | 23
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 0 | 3
Cardiac operation (Surgical and medical procedures) | 0 | 0 | 5
Dialysis (Surgical and medical procedures) | 0 | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 102
Implantable defibrillator insertion (Surgical and medical procedures) | 0 | 0 | 11
Medical device removal (Surgical and medical procedures) | 0 | 0 | 15
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 0 | 6
Surgery (Surgical and medical procedures) | 0 | 0 | 6
Vascular operation (Surgical and medical procedures) | 0 | 0 | 23
Aortic disorder (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Controlled Trial - Medtronic TAVR Systems (N=730) | Randomized Controlled Trial - SAVR (N=684) | Continued Access Study - Medtronic TAVR Systems (N=745)
Anaemia (Blood and lymphatic system disorders) | 50 | 145 | NA
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 | 40 | NA
Leukocytosis (Blood and lymphatic system disorders) | 57 | 163 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 56 | 196 | NA
Atrial Fibrillation (Cardiac disorders) | 55 | 151 | NA
Atrioventricular Block First Degree (Cardiac disorders) | 115 | 119 | NA
Bundle Branch Block Left (Cardiac disorders) | 246 | 141 | NA
Bundle Branch Block Right (Cardiac disorders) | 0 | 48 | NA
Pericardial Effusion (Cardiac disorders) | 0 | 37 | NA
Chest Pain (General disorders) | 38 | 0 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 65 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 35 | NA
Dizziness (Nervous system disorders) | 65 | 49 | NA
Acute Kidney Injury (Renal and urinary disorders) | 0 | 54 | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 69 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 42 | 0 | NA
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 109 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 39 | NA
Hypertension (Vascular disorders) | 76 | 62 | NA
Hypotension (Vascular disorders) | 0 | 41 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 60 days of receipt Medtronic (MDT) will verify presence of Confidential Information (CI) & won't censor or interfere with presentation/conclusions except to protect CI (other than Study Data) & its rights in patentable or copyrightable materials, & check technical accuracy of MDT data. If told by MDT that Publication contains CI or technical errors of MDT data, PI will make requested changes before publishing/presenting. PI will delay publication up to 90 more days, if requested.

DOCUMENTS (2):
  • Study Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT02701283/Prot_002.pdf
  • Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT02701283/SAP_003.pdf